CLINICAL TRIAL: NCT04817215
Title: A Double-Blinded, Placebo-controlled, Phase 3 Study to Evaluate the Efficacy and Safety of ORMD-0801 in Uncontrolled Type 2 DM Subjects on Diet Control Alone, Metformin Monotherapy, or Two or Three Oral Glucose-lowering Agents
Brief Title: Phase 3 Study to Evaluate the Efficacy and Safety of ORMD-0801 in Subjects With Type 2 Diabetes Mellitus
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King Hamad University Hospital, Bahrain (Other)
Collaborators: Royal College of Surgeons in Ireland - Medical University of Bahrain (Other); Oramed, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ORMD-0801-KHUH
Record Dates: First submitted 2021-03-07; First posted 2021-03-26 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — ORMD-0801

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Double-Blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients who are Drug naïve or diet controlled (Experimental)
  Interventions: Drug: ORMD-0801
- Patients on Metformin only (Experimental)
  Interventions: Drug: ORMD-0801
- Patients on two or three oral glucose-lowering agents (Experimental)
  Interventions: Drug: ORMD-0801

INTERVENTIONS:
Drug: ORMD-0801 — Randomized to receive ORMD-0801 8 mg QD or 8 mg BID or matching placebo

SUMMARY:
To compare the efficacy of ORMD-0801 to placebo in improving glycemic control as assessed by A1C in inadequately controlled T2DM subjects on diet control alone or on diet control and metformin monotherapy or two or three oral glucose-lowering agents.

To assess the safety of repeat administration of ORMD-0801 in inadequately controlled T2DM subjects on on diet control alone or on diet control and metformin monotherapy or two or three oral glucose-lowering agents.

DETAILED DESCRIPTION:
In this randomized, double-blind, double dummy, placebo-controlled study, approximately 608 eligible subjects with type 2 diabetes and inadequate control on diet control alone or on diet control and metformin monotherapy or on at least two and up to 3 oral glucose-lowering agents will undergo an initial 21-day Screening Period, followed by a 6 month Double-Blind Treatment Period and a 6 month Double-Blind Treatment Extension Period.

Screening Period:

The Investigator will review the aim of the study, study procedures and potential risks and benefits. These subjects will then sign a written informed consent during the Screening Visit 1. They will be scheduled to return to the clinic 10 days prior to randomization for Screening Visit 2. At this visit, a CGM sensor will be placed with appropriate instructions by the study team for a 10-day blinded continuous glucose monitoring (CGM) data collection by the site. Subjects will then return to the clinic after 10 days (± 1-day) for removal of the CGM sensor. The subjects will be randomized to one of the three arms of the study treatment.

6 month Double-Blind Treatment Period: After the Screening Period, subjects will be randomized to 6 months of the Double-Blind Treatment Period. In a double-blind, double dummy randomization scheme, subjects will either receive ORMD-0801 administered once-daily at night (1 x 8 mg capsule between 8 PM to 12 Midnight and no sooner than 1 hour after dinner) or ORMD-0801 8 mg (1 x 8 mg capsule) administered twice daily, each morning approximately 45 minutes (±15 minutes) prior to breakfast and each night prior to bedtime (between 8 PM to 12 Midnight and no sooner than 1 hour after dinner); or matching placebo. Subjects will receive 1 capsule approximately 45 minutes (±15 minutes) prior to breakfast and 1 capsule between 8 PM to 12 Midnight and no sooner than 1 hour after dinner.

During the Double-Blind Treatment Period commencing at Week 0 (Visit 1, CGM removal), subjects will return to the clinic every six weeks.

The visit requiring CGM application will occur 10 days prior to the CGM removal visit within ± 1-day window.

6-Month Double-Blind Treatment Extension Period: Following the completion of the Double-Blind Treatment Period, subject will enter a 6-month Double-Blind Treatment Extension Period. Subjects previously randomized to placebo during the Double-Blind Treatment Period will be randomized to receive either ORMD-0801 8 mg QD or 8 mg BID for the duration of the Double-Blind Treatment Extension Period. Subjects previously randomized to 8 mg QD or 8 mg BID during the Double-Blind Treatment Period will remain in the same treatment arm for the duration of the Double-Blind Treatment Extension Period. The Extension Period treatment assignments will remain blinded for the duration of the study.

Visits will occur at the following intervals during the 6-month Double-Blind Treatment: every six weeks. Extension Period: also every six weeks until the last visit (CGM removal and end of Double-Blind Treatment Extension Period visit).

The visit requiring CGM application will occur 10 days prior to the CGM removal visit within ± 1-day window.

All subjects completing the trial will return to the clinic in 2 weeks ± 3 days for a safety Follow-Up Visit. Subjects withdrawing prematurely from the trial will have the early termination (ET) visit procedures completed. All patients will continue to be followed in accordance with ITT principles to avoid lost to follow up and missing data.

Throughout the course of the study, subjects will measure and record fasting blood glucose levels at least 2-3 times a week [self-monitored blood glucose (SMBG)] or when they experience any symptoms of hypoglycemia using a glucose meter. Subjects will be provided a paper diary at each clinic visit and trained to record information related to fasting blood glucose and description of hypoglycemic events: time and date of occurrence; symptoms experienced, if any; treatment given, if any; and specific circumstances. Subjects will be required to bring the paper diary at each clinic visit where data will be reviewed.

Rescue Visits and Medication:

During both the Double-Blind Treatment Period and Double-Blind Treatment Extension Period, background oral glucose-lowering dose regimens will be maintained, and further dose adjustments are discouraged unless clinically indicated as follows:

Subjects will be eligible for rescue based on the following glycemic criteria:

* From Day 1 (Visit 1) through Week 6 (Visit 2), if at least two fasting SMBG levels are > 270 mg/dL in the week preceding a visit are confirmed by a single central laboratory fasting glucose > 270 mg/dL.
* From Week 6 (Visit 2) through Week 12 (Visit 3), if at least two fasting SMBG levels are > 240 mg/dL in the week preceding a visit are confirmed by a single central laboratory fasting glucose > 240 mg/dL.
* From Week 12 (Visit 3) through Week 26 (Visit 6), if at least two fasting SMBG levels are > 220 mg/dL in the week preceding a visit are confirmed by a single central laboratory fasting glucose > 220 mg/dL.
* From Week 26 (Visit 6) through the end of the study, if at least two fasting SMBG levels are > 200 mg/dL in the week preceding a visit are confirmed by a single central laboratory fasting glucose > 200 mg/dL.

Rescue will allow subjects to remain in the study, remain on double-blind study medication, complete all visits until the end of the study, and thereby, contribute to exposure and safety data. Rescue medication will be prescribed in accordance with the study Investigator's usual standard of practice.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects aged 18 - 75 years
2. Established diagnosis of T2DM for at least 6 months prior to Screening AND an A1C ≥ 7.5% but ≤ 11.0% at Screening
3. On a stable dose of at least two and up to three of the following oral glucose-lowering agents: Metformin, DPP-4 inhibitor, SGLT-2 inhibitor, thiazolidinedione, insulin secretagogue, or oral GLP-1 receptor agonists for a period of 3 months prior to Screening
4. Body mass index (BMI) of 25-40 kg/m2 at Screening and stable weight, with no more than 5 kg gain or loss in the 3 months prior to Screening
5. Renal function - eGFR ≥ 30 ml/min.
6. Females of childbearing potential must:

   1. have a negative serum pregnancy test result at Screening.
   2. agree to avoid becoming pregnant while receiving IP for at least 30 days prior to IP administration, during the entire study, and for 30 days following their last dose of IP.
   3. agree to use an acceptable method of contraception at least 30 days prior to IP administration, during the entire study, and for 30 days following their last dose of IP. Acceptable methods of contraception are hormonal contraception (contraceptive pill or injection) PLUS an additional barrier method of contraception such as a diaphragm, condom, sponge, or spermicide
   4. In the absence of hormonal contraception, double-barrier methods must be used which include a combination of any two of the following: diaphragm, condom, copper intrauterine device, sponge, or spermicide, and must be used for at least 30 days prior to administration of IP, during the entire study, and for 30 days following their last dose of IP.
   5. Abstinence (relative to heterosexual activity) can be used as the sole method of contraception if it is consistently employed as the subject's preferred and usual lifestyle and if considered acceptable by local regulatory agencies and ERCs/IRBs. Periodic abstinence (e.g., calendar, ovulation, sympto-thermal, post-ovulation methods, etc.) and withdrawal are not acceptable methods of contraception
   6. Females who are not of childbearing potential are defined as:

   i. Postmenopausal (defined as at least 12 months with no menses in women ≥45 years of age); OR ii. Have had a hysterectomy and/or bilateral oophorectomy, bilateral salpingectomy, or bilateral tubal ligation/occlusion at least 6 weeks prior to screening; OR iii. Have a congenital or acquired condition that prevents childbearing.

Exclusion Criteria:

Subjects with:

1. Type 1 diabetes
2. A history of diabetes mellitus with ketoacidosis or is assessed by the Investigator as possibly having type 1 diabetes mellitus confirmed by a C-peptide < 0.4 ng/mL (0.13 nmol/L) at Screening
3. Diabetes attributable to other secondary causes (e.g., genetic syndromes, secondary pancreatic diabetes, diabetes due to endocrinopathies, drug- or chemical-induced, and post-organ transplant).
4. Treatment involving glucosidase inhibitor, injected insulin, or injected GLP-1 receptor agonists (oral GLP-1 receptor antagonists are permitted), and pramlintide within 3 months prior to Visit 1.
5. A history of >2 episodes of severe hypoglycemia within 6 months prior to Screening.
6. A history of hypoglycemic unawareness.
7. A history of unstable angina or myocardial infarction within 6 months prior to Screening, New York Heart Association (NYHA) Grade 3 or 4 congestive heart failure (CHF), valvular heart disease, ventricular cardiac arrhythmia requiring treatment, pulmonary hypertension, cardiac surgery, coronary angioplasty, stroke or transient ischemic attack (TIA) within 6 months prior to Screening.
8. A history of uncontrolled or untreated severe hypertension defined as systolic blood pressure above or equal to 160 mmHg and/or diastolic blood pressure above or equal to 100 mmHg. A single repeat measurement will be permitted
9. Renal dysfunction: eGFR < 30 mL/min
10. A history of or active proliferative retinopathy requiring treatment
11. Psychiatric disorders that, per Investigator judgment, may have impact on the safety of the subject or interfere with subject's participation or compliance in the study
12. Laboratory abnormalities at Screening including:

    1. C-peptide < 0.4 ng/mL
    2. Abnormal serum thyrotropin (TSH) levels below the lower limit of normal or >1.5X the upper limit of normal; a single repeat test is allowable
    3. Elevated liver enzymes (alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP)) >3X the upper limit of normal; a single repeat test is allowable
    4. Very elevated fasting triglyceride levels (>600 mg/dL); a single repeat test is allowable.
    5. Any relevant abnormality that would interfere with the efficacy or the safety assessments during study treatment administration
13. Positive history of active liver disease (other than non-alcoholic hepatic steatosis), primary biliary cirrhosis, or active symptomatic gallbladder disease
14. Positive results for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), or hepatitis C virus ribonucleic acid (RNA)
15. Patient has active or history of neoplastic disease (except for adequately treated non-invasive basal cell and/or squamous cell carcinoma or carcinoma in situ of the cervix) within the past 5 years prior to baseline
16. Use of the following medications:

    1. History of use of any injectable or inhaled, basal, pre-mixed or prandial insulin (greater than 7 days) within 6 months prior to Screening
    2. Administration of thyroid preparations or thyroxine (except in subjects on stable replacement therapy) within 6 weeks prior to Screening
    3. Requirements (in the last 12 months), or may require, systemic (oral, intravenous, intramuscular) glucocorticoid therapy for more than 2 weeks during the study period. Intra-articular and/or topical corticosteroids are not considered systemic
    4. Use of medications known to modify glucose metabolism or to decrease the ability to recover from hypoglycemia such as oral, parenteral, and immunosuppressive or immunomodulating agents. Inhaled nasal steroids are permissible
17. Known allergy to soy
18. Involvement in a weight loss program and is not in the maintenance phase, or subject has started weight loss medication (e.g., orlistat or liraglutide) within 3 months prior to Screening
19. Prior bariatric surgery
20. Subject is pregnant or breast-feeding
21. Subject is a user of recreational or illicit drugs or has had a recent history (within 1 year of Screening) of drug or alcohol abuse or dependence. (Note: Alcohol abuse includes heavy alcohol intake as defined by >3 drinks per day or >14 drinks per week or binge drinking) at Screening. Occasional intermittent use of cannabinoid products will be allowed provided that no cannabinoid products have been used during the 1 week prior to each visit
22. Any condition or other factor (at the Investigator's discretion) that is deemed unsuitable for subject enrollment into the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 608 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline (Visit 1) in A1C at 26 weeks | 6 months with follow-up extension for additional six months
  • Means and mean changes from baseline over time for A1C and FPG during the Double-Blind Treatment Period and the Double-Blind Treatment Extension Period.

SECONDARY OUTCOMES:
Safety of repeat administration of ORMD-0801 in inadequately controlled T2DM subjects | 6 months with follow-up extension for additional six months
  • Safety assessed by adverse event reporting including adverse events of special interest such as hypoglycemia.

OTHER OUTCOMES:
Change from baseline (Visit 1) in CGM-parameters (using a FreeStyle Libre) | 6 months with follow-up extension for additional six months
  • Change from baseline (Visit 1) in CGM-parameters at 6 months
  o Mean Sensor Glucose, BG SD, BG CV, Time in range (TIR)-BG 70-180 mg/dL; BG 54-69 mg/dL, BG <54 mg/dL, BG 181-250 mg/dL, and BG >250 mg/dL.
Proportion of subjects achieving A1C < 8% | 6 months with follow-up extension for additional six months
  • Proportion of subjects achieving A1C < 8% at 6 months
Proportion of subjects achieving A1C < 7% | 6 months with follow-up extension for additional six months
  • Proportion of subjects achieving A1C < 7% at 6 months without reported severe hypoglycemic events.
Proportion of subjects requiring glycemic rescue therapy | 6 months with follow-up extension for additional six months
  • Proportion of subjects requiring glycemic rescue therapy and the time to rescue during the Double-Blind Treatment Period and the Double-Blind Treatment Extension Period.
Change in weight from baseline | 6 months with follow-up extension for additional six months
  • Change in weight from baseline during the Double-Blind Treatment Period and the Double-Blind Treatment Extension Period (in KG)
Means and mean changes from baseline over time for C-peptide | 6 months with follow-up extension for additional six months
  Means and mean changes from baseline over time for C-peptide during the Double-Blind Treatment Period and the Double-Blind Treatment Extension Period

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Dalal Alromaihi, Principal Investigator — King Hamad University Hospital